CLINICAL TRIAL: NCT05279989
Title: Healthy Weight and Stress Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00014499
Record Dates: First submitted 2022-02-15; First posted 2022-03-15 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Physical Disability; Obesity; Muscle Weakness; Anxiety; Depression
Keywords: Mobility impairment; Tai Chi; Stress Management; Obesity
MeSH Terms: conditions — Obesity; Muscle Weakness; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seated Tai Chi Qigong (Experimental): Participants will receive daily text messages and emails to distribute videos and record which sessions were completed. Participants can participate in 10-, 20-, or 30- min TCQ practices. Total weekly practice time will be recommended between 50-150 minutes/week (~10-30 min/day on most days). A library of existing TCQ videos will be used. All videos will demonstrate seated practice with discussions on how to accommodate mobility limitations of various types.
  Interventions: Other: Seated Tai Chi Qigong
- Control (Placebo Comparator): The control arm will receive text messages and emails with links to health information videos for the same time lengths as the intervention group. Existing video content will be reviewed and adapted to assure avoidance of topics that can impact outcome variables.
  Interventions: Other: Health Information Videos

INTERVENTIONS:
Other: Seated Tai Chi Qigong — Participants will receive seated Tai Chi Qigong videos.
  Arms: Seated Tai Chi Qigong
Other: Health Information Videos — Participants will receive videos of health information.
  Arms: Control

SUMMARY:
Approximately 1 in 10 mid-life (age 35-64) Americans have mobility impairing disabilities. People with mobility impairing disabilities are defined using the World Health Organization criteria: community living adults with mobility impairment (e.g., amputation, spinal cord injury). Women with mobility impairing disabilities often struggle with stress, abdominal fat (measured as waist circumference), lack of muscle tissue (measured as handgrip strength) and high cardiometabolic risk. This study investigates the usefulness, acceptability, and effectiveness of two strategies to reduce stress, improve health habits, reduce abdominal fat and increase muscle tissue in mid-life women with mobility impairments. These strategies involve either gentle stretching and strengthening exercises or watching informative videos.

DETAILED DESCRIPTION:
About 1 in 10 mid-life (age 35-64) Americans have mobility impairing disabilities, steadily increasing due to medical and technological innovations. People with mobility impairing disabilities (PMI) are defined using the World Health Organization criteria, as community living adults with mobility impairment (e.g., amputation, spinal cord injury). Mid-life is a critical time for people to improve their current functioning and enhance healthy aging, by improving emotional health and increasing physical activity (PA). A review showed PA improves emotional and physical health among PMI. PMI have unique challenges to meeting PA guidelines; innovative strategies are needed to achieve emotional and physical benefits for optimal health and aging.

The higher prevalence of daily stress encountered by mid-life PMI is linked to emotional health and abdominal fat (cardiometabolic disease risk) that can lead to premature mortality. This is especially so for women with mobility impairment (WMI) who have higher prevalence of excess body fat, higher cardiometabolic risk, and are not eligible for most interventions that involve PA. PA interventions also increase muscle mass, which helps to prevent cardiometabolic conditions. Although vigorous PA may not be well-suited for WMI, lighter intensity PA such as Tai Chi, Qigong and Yoga-also called meditative movement-adapted for seated practice, are a possible solution.

Tai Chi and Qigong have been tested in non-impaired populations. Our work combines these two forms of low-to-moderate PA meditative movement, Tai Chi and Qigong (TCQ), in a mind-body practice. Our research, and others', show that TCQ consistently shows strong improvement in women in depressive symptoms, anxiety, emotional eating, and sleep quality-all contributing to excess abdominal fat (measured as waist circumference), improved muscle tissue (measured as handgrip strength) and strongly associated with cardiometabolic risk. Conventional health assessment strategies do not always work well for PMI; recent innovations have yielded scalable, low-contact assessment. We have demonstrated robust recruitment, reliable questionnaire administration and strong intervention implementation expertise via social media, video sharing, and gaming platforms.

Aim 1: Assess the potential efficacy of TCQ to reduce waist circumference and increase handgrip strength compared to controls from T1 to T2 and sustain this change to T3 and T4 when compared to control.

Aim 2: Assess the potential efficacy of TCQ to reduce stress-related behaviors (depressive symptoms, anxiety, emotional eating, and sleep) that impact abdominal fat and strength when compared to control.

Aim 3: Evaluate the feasibility and acceptability of an online delivered TCQ intervention in women with mobility impairments.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling.
* Female.
* Age 35-64.
* Waist circumference >83 cm (~35 inches).
* Have a self-reported mobility impairment due to a chronic (>1 year).
* Physically disabling condition (regularly using an assistive device).
* Access to an email address and a working phone, mobile device, or personal computer or device with a high-speed internet connection.
* Understand spoken and written English and be willing to be randomized.
* Willing to engage in the intervention for 12 weeks, be available for two Zoom calls for data collection at T1, T2, T3, and T4 (Week 1, Week 4, Week 8, and Week 12).

Exclusion Criteria:

* People with full mobility.
* People who have been regularly practicing (e.g., ≥2 or more times per month for the past 6 months) any form of meditative movement including, but not limited to, Yoga, Tai Chi or Qigong.
* Pregnant, lactating, or planning to become pregnant in the next 6 months,
* Participants outside of the age range will be excluded from participation.
* Adults unable to consent and prisoners will be excluded.

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Waist Circumference assessed by measuring tape | Baseline
  Waist Circumference assessed by measuring tape
Waist Circumference assessed by measuring tape | Week 4
  Waist Circumference (cm) assessed by measuring tape
Waist Circumference measured by measuring tape | Week 8
  Waist Circumference (cm) assessed by measuring tape
Waist Circumference measured by measuring tape | Week 12
  Waist Circumference (cm) assessed by measuring tape
Handgrip strength measured by isokinetic handgrip dynamometry | Baseline
  Weight (kg) resisted measured by handgrip dynamometer
Handgrip strength measured by isokinetic handgrip dynamometry | Week 4
  Weight (kg) resisted measured by handgrip dynamometer
Handgrip strength measured by isokinetic handgrip dynamometry | Week 8
  Weight (kg) resisted measured by handgrip dynamometer
Handgrip strength measured by isokinetic handgrip dynamometry | Week 12
  Weight (kg) resisted measured by handgrip dynamometer
Depressive Symptoms assessed by Center for Epidemiologic Studies Depression Scale | Baseline
  Center for Epidemiologic Studies Depression Score ranging from 0-3, with lower scores indicating a more desirable outcome.
Depressive Symptoms assessed by Center for Epidemiologic Studies Depression Scale | Week 12
  Center for Epidemiologic Studies Depression Score ranging from 0-3, with lower scores indicating a more desirable outcome.
Anxiety assessed by Generalized Anxiety Disorder 7-item Scale | Baseline
  Generalized Anxiety Disorder 7-item Scale Score ranging from 0-21, with lower scores indicating a more desirable outcome.
Anxiety assessed by Generalized Anxiety Disorder 7-item Scale | Week 12
  Generalized Anxiety Disorder 7-item Scale Score ranging from 0-21, with lower scores indicating a more desirable outcome

SECONDARY OUTCOMES:
Emotional Eating assessed by Mindful Eating Questionnaire - 5 Factor | Baseline
  Mindful Eating Questionnaire - 5 Factor Score scored on a scale of 1-4, with higher scores signifies more mindful eating
Emotional Eating assessed by Mindful Eating Questionnaire - 5 Factor | Week 12
  Mindful Eating Questionnaire - 5 Factor Score scored on a scale of 1-4, with higher scores signifies more mindful eating
Sleep Quality assessed by the Pittsburgh Sleep Quality Index | Baseline
  Pittsburgh Sleep Quality Index Score, scored on a scale of 0-21, with higher scores indicating poorer sleep quality
Sleep Quality assessed by Pittsburgh Sleep Quality Index | Week 4
  Pittsburgh Sleep Quality Index Score, scored on a scale of 0-21, with higher scores indicating poorer sleep quality
Sleep Quality assessed by Pittsburgh Sleep Quality Index | Week 8
  Pittsburgh Sleep Quality Index Score, scored on a scale of 0-21, with higher scores indicating poorer sleep quality
Sleep Quality assessed by Pittsburgh Sleep Quality Index | Week 12
  Pittsburgh Sleep Quality Index Score, scored on a scale of 0-21, with higher scores indicating poorer sleep quality
Food Consumption Frequency assessed by the Dietary Screener Questionnaire | Baseline
  Dietary Screener Questionnaire responses measuring food consumption frequency
Food Consumption Frequency assessed by the Dietary Screener Questionnaire | Week 12
  Dietary Screener Questionnaire responses measuring food consumption frequency
Physical Functioning assessed by the Short-Form Health Survey | Baseline
  The Short-Form Health Survey Score scored 0-100, with higher scores indicating greater physical function
Physical Functioning assessed by The Short-Form Health Survey | Week 12
  The Short-Form Health Survey Score scored 0-100, with higher scores indicating greater physical function
Well-Being assessed by the Short-Form Health Survey | Baseline
  The Short-Form Health Survey Score scored 0-100, with higher scores indicating greater well-being
Well-Being assessed by the Short-Form Health Survey | Week 12
  The Short-Form Health Survey Score scored 0-100, with higher scores indicating greater well-being

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Lee, PhD, Principal Investigator — Arizona State University
Locations (1):
- Edson College of Nursing and Health Innovation, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson W, Lee C, von Schrader S. 2017 disability status report: United states. In: Ithaca, NY: Cornell University Yang-Tan Institute on Employment and Disability (YTI); 2019
- [Background] Kraus L, Lauer E, Coleman R, Houtenville A. 2017 disability statistics annual report. Durham, NH: University of New Hampshire; 2018.
- [Background] Brault M. Americans with disabilities: 2005. In. Current Populations Reports. Washington, DC: US Census Bureau; 2008:70-117.
- [Background] Institute of Medicine (US) Committee on Disability in America; Field MJ, Jette AM, editors. The Future of Disability in America. Washington (DC): National Academies Press (US); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK11434/ PMID 20669428
- [Background] UN World Health Organization (WHO). World report on disability : Summary, 2011, who/nmh/vip/11.01. https://www.refworld.org/docid/50854a322.html. Published 2011. Accessed Feburary 1, 2021.
- [Background] World Health Organization. International statistical classification of diseases and related health problems (icd-10). 10th ed. Geneva, Switzerland: World Health Organization; 1992.
- [Background] World Health Organization. Health topics: Disability. https://www.who.int/health-topics/disability#tab=tab_1. Published 2021. Accessed February 1, 2021.
- [Background] Karvonen-Gutierrez CA. The importance of disability as a health issue for mid-life women. Womens Midlife Health. 2015 Oct 14;1:10. doi: 10.1186/s40695-015-0011-x. eCollection 2015. PMID 30766697
- [Background] Selph SS, Skelly AC, Wasson N, Dettori JR, Brodt ED, Ensrud E, Elliot D, Dissinger KM, Hart E, Kantner S, Graham E, Junge M, Dana T, McDonagh M. Physical Activity and the Health of Wheelchair Users: A Systematic Review in Multiple Sclerosis, Cerebral Palsy, and Spinal Cord Injury [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2021 Oct. Report No.: 21(22)-EHC017. Available from http://www.ncbi.nlm.nih.gov/books/NBK574873/ PMID 34723448
- [Background] Nosek MA, Hughes RB, Robinson-Whelen S, Taylor HB, Howland CA. Physical activity and nutritional behaviors of women with physical disabilities: physical, psychological, social, and environmental influences. Womens Health Issues. 2006 Nov-Dec;16(6):323-33. doi: 10.1016/j.whi.2006.08.002. PMID 17188215
- [Background] Rosenberg DE, Bombardier CH, Hoffman JM, Belza B. Physical activity among persons aging with mobility disabilities: shaping a research agenda. J Aging Res. 2011;2011:708510. doi: 10.4061/2011/708510. Epub 2011 Jun 26. PMID 21748010
- [Background] Froehlich-Grobe K, Lee J, Washburn RA. Disparities in obesity and related conditions among Americans with disabilities. Am J Prev Med. 2013 Jul;45(1):83-90. doi: 10.1016/j.amepre.2013.02.021. PMID 23790992
- [Background] Harris RB, Zhou J, Youngblood BD, Rybkin II, Smagin GN, Ryan DH. Effect of repeated stress on body weight and body composition of rats fed low- and high-fat diets. Am J Physiol. 1998 Dec;275(6):R1928-38. doi: 10.1152/ajpregu.1998.275.6.R1928. PMID 9843882
- [Background] Hughes RB, Nosek MA, Robinson-Whelen S. Correlates of depression in rural women with physical disabilities. J Obstet Gynecol Neonatal Nurs. 2007 Jan-Feb;36(1):105-114. doi: 10.1111/j.1552-6909.2006.00122.x. PMID 17238955
- [Background] Hughes RB, Robinson-Whelen S, Taylor HB, Hall JW. Stress self-management: an intervention for women with physical disabilities. Womens Health Issues. 2006 Nov-Dec;16(6):389-99. doi: 10.1016/j.whi.2006.08.003. PMID 17188222
- [Background] Morgan RO, Byrne MM, Hughes RB, Petersen NJ, Taylor HB, Robinson-Whelen S, Hasche JC, Nosek MA. Do secondary conditions explain the relationship between depression and health care cost in women with physical disabilities? Arch Phys Med Rehabil. 2008 Oct;89(10):1880-6. doi: 10.1016/j.apmr.2008.03.011. PMID 18929016
- [Background] Nosek MA, Hughes RB, Petersen NJ, Taylor HB, Robinson-Whelen S, Byrne M, Morgan R. Secondary conditions in a community-based sample of women with physical disabilities over a 1-year period. Arch Phys Med Rehabil. 2006 Mar;87(3):320-7. doi: 10.1016/j.apmr.2005.11.003. PMID 16500164
- [Background] Nosek MA, Hughes RB, Robinson-Whelen S. The complex array of antecedents of depression in women with physical disabilities: implications for clinicians. Disabil Rehabil. 2008;30(3):174-83. doi: 10.1080/09638280701532219. PMID 17852240
- [Background] Nosek MA, Robinson-Whelen S, Hughes RB, Nosek TM. An Internet-based virtual reality intervention for enhancing self-esteem in women with disabilities: Results of a feasibility study. Rehabil Psychol. 2016 Nov;61(4):358-370. doi: 10.1037/rep0000107. Epub 2016 Oct 6. PMID 27709978
- [Background] Nosek MA, Robinson-Whelen S, Hughes RB, Petersen NJ, Taylor HB, Byrne MM, Morgan R. Overweight and obesity in women with physical disabilities: associations with demographic and disability characteristics and secondary conditions. Disabil Health J. 2008 Apr;1(2):89-98. doi: 10.1016/j.dhjo.2008.01.003. PMID 21122716
- [Background] Robinson-Whelen S, Hughes RB, Taylor HB, Colvard M, Mastel-Smith B, Nosek MA. Improving the health and health behaviors of women aging with physical disabilities: A peer-led health promotion program. Womens Health Issues. 2006 Nov-Dec;16(6):334-45. doi: 10.1016/j.whi.2006.05.002. PMID 17188216
- [Background] Robinson-Whelen S, Hughes RB, Taylor HB, Hall JW, Rehm LP. Depression self-management program for rural women with physical disabilities. Rehabil Psychol. 2007;52(3):254-262.
- [Background] Robinson-Whelen S, Hughes RB, Taylor HB, Markley R, Vega JC, Nosek TM, Nosek MA. Promoting psychological health in women with SCI: Development of an online self-esteem intervention. Disabil Health J. 2020 Apr;13(2):100867. doi: 10.1016/j.dhjo.2019.100867. Epub 2019 Nov 7. PMID 31757776
- [Background] Robinson-Whelen S, Taylor HB, Hughes RB, Nosek MA. Depressive symptoms in women with physical disabilities: identifying correlates to inform practice. Arch Phys Med Rehabil. 2013 Dec;94(12):2410-2416. doi: 10.1016/j.apmr.2013.07.013. Epub 2013 Jul 31. PMID 23911557
- [Background] Robinson-Whelen S, Taylor HB, Hughes RB, Wenzel L, Nosek MA. Depression and depression treatment in women with spinal cord injury. Top Spinal Cord Inj Rehabil. 2014 Winter;20(1):23-31. doi: 10.1310/sci2001-23. PMID 24574819
- [Background] Stefanaki C, Pervanidou P, Boschiero D, Chrousos GP. Chronic stress and body composition disorders: implications for health and disease. Hormones (Athens). 2018 Mar;17(1):33-43. doi: 10.1007/s42000-018-0023-7. Epub 2018 Apr 27. PMID 29858868
- [Background] Nosek MA, Robinson-Whelen S, Ledoux TA, Hughes RB, O'Connor DP, Lee RE, Goe R, Silveira SL, Markley R, Nosek TM; GoWoman Consortium. A pilot test of the GoWoman weight management intervention for women with mobility impairments in the online virtual world of Second Life(R). Disabil Rehabil. 2019 Nov;41(22):2718-2729. doi: 10.1080/09638288.2018.1473511. Epub 2018 Jun 11. PMID 29889580
- [Background] Lu EY, Lee P, Cai S, So WWY, Ng BFL, Jensen MP, Cheung WM, Tsang HWH. Qigong for the treatment of depressive symptoms: Preliminary evidence of neurobiological mechanisms. Int J Geriatr Psychiatry. 2020 Nov;35(11):1393-1401. doi: 10.1002/gps.5380. Epub 2020 Aug 6. PMID 32662069
- [Background] Zou L, Sasaki JE, Wei GX, Huang T, Yeung AS, Neto OB, Chen KW, Hui SS. Effects of Mind(-)Body Exercises (Tai Chi/Yoga) on Heart Rate Variability Parameters and Perceived Stress: A Systematic Review with Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2018 Oct 31;7(11):404. doi: 10.3390/jcm7110404. PMID 30384420
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Coker J, Cuthbert J, Ketchum JM, Holicky R, Huston T, Charlifue S. Re-inventing yourself after spinal cord injury: a site-specific randomized clinical trial. Spinal Cord. 2019 Apr;57(4):282-292. doi: 10.1038/s41393-018-0230-8. Epub 2018 Dec 20. PMID 30573769
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Terrill AL, Hartoonian N, Beier M, Salem R, Alschuler K. The 7-item generalized anxiety disorder scale as a tool for measuring generalized anxiety in multiple sclerosis. Int J MS Care. 2015 Mar-Apr;17(2):49-56. doi: 10.7224/1537-2073.2014-008. PMID 25892974
- [Background] Randpack: Randomization routines for clinical trials, r package [computer program]. Version 1.3.5: Bioconductor; 2018.
- [Background] Zhou Y, Wang Q, Larkey L, James D, Cui H. Tai Chi Effects on Heart Rate Variability: A Systematic Review and Meta-Analysis. J Integr Complement Med. 2024 Feb;30(2):121-132. doi: 10.1089/jicm.2022.0682. Epub 2023 Sep 11. PMID 37695835
- [Background] Larkey LK, James D, Belyea M, Jeong M, Smith LL. Body Composition Outcomes of Tai Chi and Qigong Practice: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Int J Behav Med. 2018 Oct;25(5):487-501. doi: 10.1007/s12529-018-9725-0. PMID 29856007
- [Background] Yin J, Dishman RK. The effect of tai chi and qigong practice on depression and anxiety symptoms: A systematic review and meta-regression analysis of randomized controlled trials. Ment Health Phys Act. 2014;7(3):135-146.
- [Background] Zeng Y, Luo T, Xie H, Huang M, Cheng AS. Health benefits of qigong or tai chi for cancer patients: a systematic review and meta-analyses. Complement Ther Med. 2014 Feb;22(1):173-86. doi: 10.1016/j.ctim.2013.11.010. Epub 2013 Dec 18. PMID 24559833
- [Background] Qi Y, Zhang X, Zhao Y, Xie H, Shen X, Niu W, Wang Y. The effect of wheelchair Tai Chi on balance control and quality of life among survivors of spinal cord injuries: A randomized controlled trial. Complement Ther Clin Pract. 2018 Nov;33:7-11. doi: 10.1016/j.ctcp.2018.07.004. Epub 2018 Jul 20. PMID 30396629
- [Background] Tsang WW, Gao KL, Chan KM, Purves S, Macfarlane DJ, Fong SS. Sitting tai chi improves the balance control and muscle strength of community-dwelling persons with spinal cord injuries: a pilot study. Evid Based Complement Alternat Med. 2015;2015:523852. doi: 10.1155/2015/523852. Epub 2015 Jan 21. PMID 25688276
- [Background] Lee RE, O'Neal A, Cameron C, Hughes RB, O'Connor DP, Ohri-Vachaspati P, Todd M, Nosek MA. Developing Content for the Food Environment Assessment Survey Tool (FEAST): A Systematic Mixed Methods Study with People with Disabilities. Int J Environ Res Public Health. 2020 Oct 24;17(21):7781. doi: 10.3390/ijerph17217781. PMID 33114296
- [Background] Aschner P, Buendia R, Brajkovich I, Gonzalez A, Figueredo R, Juarez XE, Uriza F, Gomez AM, Ponte CI. Determination of the cutoff point for waist circumference that establishes the presence of abdominal obesity in Latin American men and women. Diabetes Res Clin Pract. 2011 Aug;93(2):243-247. doi: 10.1016/j.diabres.2011.05.002. Epub 2011 May 31. PMID 21632141
- [Background] Zhu S, Heymsfield SB, Toyoshima H, Wang Z, Pietrobelli A, Heshka S. Race-ethnicity-specific waist circumference cutoffs for identifying cardiovascular disease risk factors. Am J Clin Nutr. 2005 Feb;81(2):409-15. doi: 10.1093/ajcn.81.2.409. PMID 15699228
- [Background] Pocock SJ, Simon R. Sequential treatment assignment with balancing for prognostic factors in the controlled clinical trial. Biometrics. 1975 Mar;31(1):103-15. PMID 1100130
- [Background] Chen SC, Ueng KC, Lee SH, Sun KT, Lee MC. Effect of t'ai chi exercise on biochemical profiles and oxidative stress indicators in obese patients with type 2 diabetes. J Altern Complement Med. 2010 Nov;16(11):1153-9. doi: 10.1089/acm.2009.0560. Epub 2010 Oct 25. PMID 20973735
- [Background] Cheung BM, Lo JL, Fong DY, Chan MY, Wong SH, Wong VC, Lam KS, Lau CP, Karlberg JP. Randomised controlled trial of qigong in the treatment of mild essential hypertension. J Hum Hypertens. 2005 Sep;19(9):697-704. doi: 10.1038/sj.jhh.1001884. PMID 15905884
- [Background] Hui SS, Xie YJ, Woo J, Kwok TC. Practicing Tai Chi had lower energy metabolism than walking but similar health benefits in terms of aerobic fitness, resting energy expenditure, body composition and self-perceived physical health. Complement Ther Med. 2016 Aug;27:43-50. doi: 10.1016/j.ctim.2016.05.006. Epub 2016 May 20. PMID 27515875
- [Background] Hung HM, Yeh SH, Chen CH. Effects of Qigong Exercise on Biomarkers and Mental and Physical Health in Adults With at Least One Risk Factor for Coronary Artery Disease. Biol Res Nurs. 2016 May;18(3):264-73. doi: 10.1177/1099800415617017. Epub 2015 Nov 20. PMID 26590130
- [Background] Framson C, Kristal AR, Schenk JM, Littman AJ, Zeliadt S, Benitez D. Development and validation of the mindful eating questionnaire. J Am Diet Assoc. 2009 Aug;109(8):1439-44. doi: 10.1016/j.jada.2009.05.006. PMID 19631053
- [Background] Monk TH, Reynolds CF, Kupfer DJ, Buysse DJ, Coble PA, Hayes AJ, MacHen MA, Petrie SR, Ritenour AM. The Pittsburgh Sleep Diary. J Sleep Res. 1994 Jun;3(2):111-120. PMID 10607115